CLINICAL TRIAL: NCT00659022
Title: Accelerated Growth of Synchronous Colorectal Liver Metastases: Effects of Neo-adjuvant Therapy
Brief Title: Neo-adjuvant Therapy and the Effect on Synchronous Metastatic Growth
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: T.J.M Ruers, PhD, The Netherlands Cancer Institute/ Antoni van Leeuwenhoek Hospital Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SILENT
Record Dates: First submitted 2008-04-03; First posted 2008-04-16 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Neoplasms; Liver Neoplasms
Keywords: colorectal cancer; liver metastases; angiogenesis; metabolism
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms | interventions — Bevacizumab; Neoadjuvant Therapy; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): immediate surgery of the primary colorectal tumor, no neoadjuvant therapy
  Interventions: Procedure: immediate surgery (resection of primary colorectal tumor)
- B (Experimental): neoadjuvant treatment with bevacizumab during 7 weeks prior to surgery of the colorectal primary
  Interventions: Drug: neo-adjuvant treatment with bevacizumab
- C (Experimental): neoadjuvant treatment with CAPOX during 7 weeks prior to surgery of the colorectal primary
  Interventions: Drug: neoadjuvant treatment with capecitabine and oxaliplatin
- D (Experimental): neoadjuvant treatment with bevacizumab and CAPOX during 7 weeks prior to surgery of the colorectal primary
  Interventions: Drug: neo-adjuvant treatment with bevacizumab, capecitabine and oxaliplatin

INTERVENTIONS:
Procedure: immediate surgery (resection of primary colorectal tumor) — no neo-adjuvant treatment, immediate surgery
  Arms: A
Drug: neo-adjuvant treatment with bevacizumab — neoadjuvant treatment with bevacizumab during 7 weeks prior to surgery of the colorectal primary
  Other Names: Avastin
  Arms: B
Drug: neoadjuvant treatment with capecitabine and oxaliplatin — neoadjuvant treatment with CAPOX during 7 weeks prior to surgery of the colorectal primary
  Other Names: Xeloda; Eloxatin
  Arms: C
Drug: neo-adjuvant treatment with bevacizumab, capecitabine and oxaliplatin — neoadjuvant treatment with bevacizumab and CAPOX during 7 weeks prior to surgery of the colorectal primary
  Other Names: Avastin; Xeloda; Eloxatin
  Arms: D

SUMMARY:
Study Hypothesis

• As well as in animal models as in patients with colorectal cancer resection of the primary tumor resulted in increase in vascular density, metabolism and secondary tumor growth of the distant metastases. These data strongly suggest an inhibitory effect of the primary tumor on the outgrowth of its metastases.

In this study we investigate whether pre-operative treatment with the anti-angiogenic agent bevacizumab and/or chemotherapy before resection of the primary colorectal tumor shifts the balance between angiogenic and anti-angiogenic factors in favor of the anti-angiogenic factors and results in reduced growth of the liver metastases.

Eligibility

* Histological proven colorectal cancer without signs of bowel obstruction or bleeding
* Synchronous liver metastases
* WHO performance status 0-1

Treatment

* Arm A: immediate surgery of the primary colorectal tumor, no neoadjuvant therapy
* Arm B: neoadjuvant treatment with bevacizumab during 7 weeks prior to surgery of the colorectal primary
* Arm C: neoadjuvant treatment with CAPOX during 7 weeks prior to surgery of the colorectal primary
* Arm D: neoadjuvant treatment with bevacizumab and CAPOX during 7 weeks prior to surgery of the colorectal primary

Primary endpoint Difference in response of liver metastases to resection of the primary tumor between the experimental groups and the control group, as determined by histopathological scoring of vascular density, apoptotic and mitotic index and by measurement of the metabolic activity of liver metastases by FDG-PET and SUV measurements.

Secondary endpoints Toxicity of neo-adjuvant treatment Complications of surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven primary colorectal cancer and synchronous unresectable liver metastases with or without additional extrahepatic disease (primary tumor in situ). Unresectable liver metastases defined as too extensive hepatic involvement or extrahepatic disease.
* Measurable liver metastases on CT scan (RECIST), positive signal of liver metastases on FDG-PET scan
* Age: 18-80 years
* WHO performance scale 0-1
* ASA category I or II
* Negative pregnancy test in women with childbearing potential
* Life expectancy > 12 weeks
* Laboratory values obtained ≤ 3 weeks prior to study entry, disease evaluation performed ≤ 3 weeks prior to study entry. Adequate bone marrow function (Hb > 6.5 mmol/L, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L), renal function (serum creatinine < 1.5 x ULN or creatinine clearance ≥ 50 mL/min (calculated according to Cockroft and Gault), liver function (ASAT and ALAT ≤ 3 x upper normal limit, serum bilirubin ≤ 2 x upper normal limit)
* Written informed consent

Exclusion Criteria:

* Signs of bowel obstruction or bleeding from primary tumor
* Prior chemotherapy treatment for advanced disease, prior treatment with anti-angiogenic drugs
* Resectable liver metastases
* Diabetes mellitus
* Continuous use of immunosuppressive agents
* Pregnancy or lactation
* Contra-indications for systemic therapy with bevacizumab (Avastin)/ chemotherapy (Xelox)
* Concurrent severe or uncontrolled disease (i.e. uncontrolled hypertension, congestive heart failure, myocardial infarction < 12 months, chronic active infection)
* Sensory neuropathy > grade 1
* Serious non-healing wound or ulcer
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measures
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to start of bevacizumab
* Bleeding disorders or coagulopathy or need for full-dose anticoagulation
* Signs or symptoms of brain metastases
* Cerebrovascular accident or transient ischemic attack within the past 12 months
* Impairment of gastrointestinal function or -disease that may significantly impair the absorption of oral drugs (i.e. uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow tablets)
* Presence of proteinuria at baseline as defined by: patients with > 1 g of protein/24 hr by a 24-hour urine collection.
* Any concomitant disorder preventing the safe administration of study drugs or surgical procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Difference in response of liver metastases between control group and experimental groups determined by histopathological scoring of vascular density,apoptotic and mitotic index | 12 weeks
Difference in response of liver metastases between control group and experimental groups determined by FDG-PET | 12 weeks

SECONDARY OUTCOMES:
Toxicity of neo-adjuvant treatment | 12 weeks
Complications of surgery | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, PhD, Principal Investigator — The Netherlands Cancer Institute; Kees Punt, PhD, Principal Investigator — Radboud University Nijmegen Medical Center; Wim Oyen, PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (2):
- Netherlands (2):
  - The Netherlands Cancer Institute/ Antoni van Leeuwenhoek Hospital, Amsterdam
  - Radboud University Nijmegen Medical Center, Nijmegen

REFERENCES:
- [Background] Gorelik E, Segal S, Feldman M. On the mechanism of tumor "concomitant immunity". Int J Cancer. 1981 Jun 15;27(6):847-56. doi: 10.1002/ijc.2910270618. No abstract available. PMID 7287231
- [Background] O'Reilly MS, Holmgren L, Shing Y, Chen C, Rosenthal RA, Moses M, Lane WS, Cao Y, Sage EH, Folkman J. Angiostatin: a novel angiogenesis inhibitor that mediates the suppression of metastases by a Lewis lung carcinoma. Cell. 1994 Oct 21;79(2):315-28. doi: 10.1016/0092-8674(94)90200-3. PMID 7525077
- [Background] O'Reilly MS, Boehm T, Shing Y, Fukai N, Vasios G, Lane WS, Flynn E, Birkhead JR, Olsen BR, Folkman J. Endostatin: an endogenous inhibitor of angiogenesis and tumor growth. Cell. 1997 Jan 24;88(2):277-85. doi: 10.1016/s0092-8674(00)81848-6. PMID 9008168
- [Background] Peeters CF, Westphal JR, de Waal RM, Ruiter DJ, Wobbes T, Ruers TJ. Vascular density in colorectal liver metastases increases after removal of the primary tumor in human cancer patients. Int J Cancer. 2004 Nov 20;112(4):554-9. doi: 10.1002/ijc.20374. PMID 15382035
- [Background] Yang AD, Bauer TW, Camp ER, Somcio R, Liu W, Fan F, Ellis LM. Improving delivery of antineoplastic agents with anti-vascular endothelial growth factor therapy. Cancer. 2005 Apr 15;103(8):1561-70. doi: 10.1002/cncr.20942. PMID 15754332
- [Background] Heldin CH, Rubin K, Pietras K, Ostman A. High interstitial fluid pressure - an obstacle in cancer therapy. Nat Rev Cancer. 2004 Oct;4(10):806-13. doi: 10.1038/nrc1456. PMID 15510161
- [Background] Tong RT, Boucher Y, Kozin SV, Winkler F, Hicklin DJ, Jain RK. Vascular normalization by vascular endothelial growth factor receptor 2 blockade induces a pressure gradient across the vasculature and improves drug penetration in tumors. Cancer Res. 2004 Jun 1;64(11):3731-6. doi: 10.1158/0008-5472.CAN-04-0074. PMID 15172975
- [Background] Jain RK. Normalization of tumor vasculature: an emerging concept in antiangiogenic therapy. Science. 2005 Jan 7;307(5706):58-62. doi: 10.1126/science.1104819. PMID 15637262